CLINICAL TRIAL: NCT01101698
Title: Influence of Vitamin K2 Administration on Vessel Calcification Markers in Patients With Chronic Kidney Disease
Brief Title: Vitamin K2 and Vessel Calcification in Chronic Kidney Disease Patients
Acronym: CACSK2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Prof Michał Nowicki, Department of Nephrology, Hypertensiology and Kidney Transplantation Medical University of Łódź
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CACSK2
Record Dates: First submitted 2010-04-09; First posted 2010-04-12 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Kidney Diseases; Coronary Artery Calcification
Keywords: Vitamin K; chronic kidney disease; coronary artery calcification; intima media thickness
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin K2, calcification score changes, vitamin D (Active Comparator): 90 μg vitamin K2+10μg cholecalciferol
  Interventions: Drug: Vitamin K2+10μg cholecalciferol; Drug: Vitamin D
- Vitamin D, calcium score changes (Active Comparator): 10μg cholecalciferol (vitamin D)
  Interventions: Drug: Vitamin K2+10μg cholecalciferol

INTERVENTIONS:
Drug: Vitamin K2+10μg cholecalciferol — Pills of: 90 μg vitamin K2+10μg cholecalciferol once daily during 9 months
Drug: Vitamin D — Pills of: 10μg cholecalciferol (Vitamin D)once daily during 9 months
  Arms: Vitamin K2, calcification score changes, vitamin D

SUMMARY:
Vessel calcification is a recognised cardiovascular morbidity risk factor in patients with chronic kidney disease (CKD). Recent reports indicate a significant role of Matrix Gla-protein (MGP) in decreasing calcification processes. MGP is excretion protein whose mechanism of action is not yet fully explained and which to be activated requires phosphorylation and carboxylation where cofactor is vitamin K. These observations indicate that shortage of vitamin K is a significant risk factor for the development of vessel calcification. Another calcification risk factor in CKD patients are calcium-phosphate disturbances and insufficiency of vitamin D3 which in physiological concentration stimulates MGP transcription. The aim of this study is estimation of influence of vitamin K2 administration over the period of 9 months on vessel calcification in 3.- 5. stage CKD patients.

It is a prospective, randomised double-blind study carried out in parallel groups. 60 patients with CKD (GFR 15-60 ml/min) with calcium score >10 (Agatston scoring system) will be qualified for the study. On the basis of randomised selection, patients will be divided into two groups: 30 patients will be given 90 μg vitamin K2 + 10 μg and cholecalciferol 30 patients will be given only 10 μg cholecalciferol. After a 9-month treatment the image diagnostic will be carried out in order to estimate the degree of vessel calcification.

DETAILED DESCRIPTION:
Vessel calcification is a recognised cardiovascular morbidity risk factor in patients with chronic kidney disease (CKD). Recent reports indicate a significant role of Matrix Gla-protein (MGP) in decreasing calcification processes. MGP is excretion protein whose mechanism of action is not yet fully explained and which to be activated requires phosphorylation and carboxylation where cofactor is vitamin K. Immunohistochemical tests showed a high level of un-carboxylated MGP in calcified vessels. These observations indicate that shortage of vitamin K is a significant risk factor for the development of vessel calcification. On the other hand CKD patients often display shortages of this vitamin. Another calcification risk factor in CKD patients are calcium-phosphate disturbances and insufficiency of vitamin D3 which in physiological concentration stimulates MGP transcription. Cranenburg et al. showed a decrease vessel calcification in dialysis patients treated with vitamin K2. Vitamin K2 exists in two forms K1 and K2, however only the K2 form displays calcification decreasing properties. There are currently no similar studies in patients with chronic kidney disease who do not require renal replacement therapy.

The aim of study. The aim of this study is estimation of influence of vitamin K2 administration over the period of 9 months on vessel calcification in 3.- 5. stage CKD patients.

Materials and methods. It is a prospective, randomised double-blind study carried out in parallel groups. 60 patients with CKD (GFR 15-60 ml/min) whose renal replacement therapy is to commence not earlier than in 9 months are planned to be qualified for the study. After familiarizing the patients with the aims of the study and obtaining their written consent, non-invasive tests will be carried out in order to estimate the presence and degree of vessel calcification: common carotid artery intima media thickness (CCA-IMT) by ultrasound examination, coronary artery calcium score (CACS) by multiscan CT as well as the presence of calcified heart valves by ultrasound examination. Patients with calcium score >10 (Agatston scoring system) will be qualified for the study. On the basis of randomised selection, patients will be divided into two groups: 30 patients will be given 90 μg vitamin K2+10 μg cholecalciferol (Vitamin D)and 30 patients will be given only 10 μg cholecalciferol. After a 9-month treatment the image diagnostic will be carried out in order to estimate the degree of vessel calcification. Patients and their basic laboratory test will be evaluated during the study period by a nephrologists on a monthly basis. First, at the commencement of the study, then after 3, 6 and finally after 9 months during the last visit, 10 ml of serum and plasma will be taken and frozen in order to conduct special marking tests: phosphorylated MGP (pMGP), uncarboxylated MGP (ucMGP), 25-OH cholecalciferol, hsCRP.

Scheduling Study Visits:

Visit 0 Screening Period

1. Review of inclusion and exclusion criteria
2. Obtain informed consent
3. Obtain weight and height
4. Obtain CACS, CCA-IMT
5. Obtain heart ultrasonography
6. Review concomitant therapy

Visit 1 - Randomization

1. Review of inclusion and exclusion criteria
2. Medical history for concomitant disorders (hypertension, heart ischemic diseases, diabetes mellitus)
3. Collect blood for serum chemistry (creatinine, albumin, intact PTH, calcium, phosphor, uric acid, lipids, glucose, kaolin-kephalin time, prothrombin index and blood morphology.
4. Collect blood for pMGP, ucMGP, 25-OH cholecalciferol, hsCRP
5. Review concomitant therapy
6. Randomization to: 90 μg vitamin K2+10μg cholecalciferol or 10μg cholecalciferol (Vitamin D) during 9 months

Visit 2,4,5,7,8 Visits every month

1. Complete physical examination
2. GFR obtain
3. Drug dispension

Visit 3,6 and after 9 months:

1. Complete physical examination
2. GFR obtain
3. Collect blood for serum chemistry (creatinine, albumin, intact PTH, calcium, phosphor, uric acid, lipids, glucose, kaolin-kephalin time, prothrombin index and blood morphology.
4. Collect blood for pMGP, ucMGP, 25-OH cholecalciferol, hsCRP
5. Obtain CACS, CCA-IMT
6. Obtain heart ultrasonography
7. Review concomitant therapy

ELIGIBILITY:
Inclusion Criteria:

1. Subject with chronic kidney disease (creatinine clearance 15-60 ml/min/1,73m2 by Cockroft-Gault formula)
2. Patient has a life without dialysis therapy of more than 9 months
3. Subject in 30-70 years of age
4. Calcium score >10 (as per Agatston scoring system)

Exclusion Criteria:

1. Atherosclerosis generalisata (myocardial infarction treated with PTCA - Percutaneous Transluminal Coronary Angioplasty or CABG - Coronary Artery Bypass Graft, symptomatic heart insufficiency, cerebrovascular accident)
2. Subject with a history of cardiac abnormalities, including symptomatic or asymptomatic arrhythmias (atrial fibrillation)
3. Patient with cardiac pacemaker
4. Subject requires long-term use of vitamin K antagonists

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Changes in coronary artery calcification score | 9 months

SECONDARY OUTCOMES:
Changes in common carotid artery intima media thickness | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology, Hypertension and Kidney Transplantation, Lodz, Poland

REFERENCES:
- [Background] Pilkey RM, Morton AR, Boffa MB, Noordhof C, Day AG, Su Y, Miller LM, Koschinsky ML, Booth SL. Subclinical vitamin K deficiency in hemodialysis patients. Am J Kidney Dis. 2007 Mar;49(3):432-9. doi: 10.1053/j.ajkd.2006.11.041. PMID 17336705
- [Background] Schurgers LJ, Cranenburg EC, Vermeer C. Matrix Gla-protein: the calcification inhibitor in need of vitamin K. Thromb Haemost. 2008 Oct;100(4):593-603. PMID 18841280
- [Background] Cranenburg EC, Vermeer C, Koos R, Boumans ML, Hackeng TM, Bouwman FG, Kwaijtaal M, Brandenburg VM, Ketteler M, Schurgers LJ. The circulating inactive form of matrix Gla Protein (ucMGP) as a biomarker for cardiovascular calcification. J Vasc Res. 2008;45(5):427-36. doi: 10.1159/000124863. Epub 2008 Apr 10. PMID 18401181
- [Derived] Kurnatowska I, Grzelak P, Masajtis-Zagajewska A, Kaczmarska M, Stefanczyk L, Vermeer C, Maresz K, Nowicki M. Effect of vitamin K2 on progression of atherosclerosis and vascular calcification in nondialyzed patients with chronic kidney disease stages 3-5. Pol Arch Med Wewn. 2015;125(9):631-40. doi: 10.20452/pamw.3041. Epub 2015 Jul 15. PMID 26176325